CLINICAL TRIAL: NCT04780984
Title: A Phase 2, Randomized, Partially-blinded, Parallel Group, Dose-ranging Study to Assess the Pharmacodynamics, Relative Bioavailability, and Safety of of Tiotropium Bromide Inhalation Solution in Subjects With COPD
Brief Title: Tiotropium Bromide Inhalation Solution in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nephron Pharmaceuticals Corporation (Industry)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neph-0002
Record Dates: First submitted 2020-11-02; First posted 2021-03-04 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo, 2mL
  Interventions: Drug: Placebo
- Group 1 Tiotropium Bromide Inhalation Solution (Experimental): Treatment Dose (µg) Volume (mL) Concentration (µg/mL)
  8 µg, 2.0 mL, 4 µg/mL
  Interventions: Drug: Tiotropium bromide inhalation solution
- Group 2 Tiotropium Bromide Inhalation Solution (Experimental): Treatment Dose (µg) Volume (mL) Concentration (µg/mL)
  16 µg, 2.0 mL, 8 µg/mL
  Interventions: Drug: Tiotropium bromide inhalation solution
- Group 3 Tiotropium Bromide Inhalation Solution (Experimental): Treatment Dose (µg) Volume (mL) Concentration (µg/mL)
  24 µg, 2.0 mL, 12 µg/mL
  Interventions: Drug: Tiotropium bromide inhalation solution
- Spiriva Respimat (Active Comparator): 5 ug, 2 actuations, 2.5 µg/actuation
  Interventions: Drug: Tiotropium bromide inhalation solution

INTERVENTIONS:
Drug: Tiotropium bromide inhalation solution — Tiotropium bromide inhalation solution
  Arms: Group 1 Tiotropium Bromide Inhalation Solution; Group 2 Tiotropium Bromide Inhalation Solution; Group 3 Tiotropium Bromide Inhalation Solution; Spiriva Respimat
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
A Phase 2, Randomized, Partially-blinded, Parallel Group, Dose-ranging Study to Assess the Pharmacodynamics, Relative Bioavailability, and Safety of Three Doses of Tiotropium Bromide Inhalation Solution in Subjects with Chronic Obstructive Pulmonary Disease

DETAILED DESCRIPTION:
Objectives:

Primary:

• To determine the effect of once daily dosing with tiotropium bromide inhalation solution for 22 consecutive days on trough forced expiratory volume in 1 second (FEV1) change from baseline compared with that of placebo inhalation solution in subjects with chronic obstructive pulmonary disease (COPD).

Secondary:

* To determine the effect of once daily dosing with tiotropium bromide inhalation solution for 22 consecutive days on trough FEV1 change from baseline compared with that of Spiriva Respimat; area under the curve (AUC) FEV10-6 change from baseline compared with that of placebo and Spiriva Respimat; and trough forced vital capacity (FVC) change from baseline compared with that of placebo and Spiriva Respimat
* To assess the safety and tolerability of tiotropium bromide inhalation solution in subjects with COPD
* To assess the relative bioavailability of tiotrop

ELIGIBILITY:
Inclusion Criteria:

* Males and nonpregnant females, ages 40 to 80 years old, inclusive.
* On a stable COPD medication regimen defined as: no new medications for or changes to medications (dose/frequency) used to manage COPD within 60 days of screening.
* Willing and able to give informed consent and follow all study procedures and requirements.
* Body mass index <35.
* Female subjects of child-bearing potential1 who are non-lactating, are using and agree tocontinue using an acceptable method of contraception for at least 4 weeks prior to first dose of study drug and until 12 weeks after last dose, and have a negative serum pregnancy test during screening. Adequate contraception is defined as a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label, for example: abstinence from penile-vaginal intercourse; oral contraceptives, either combined or progestogen alone; injectable progestogen; implants of etonogestrel or levonorgestrel; estrogenic vaginal ring; percutaneous contraceptive patches; intrauterine device or intrauterine system; male partner sterilization at least 6 months prior to the female subject's screening visit, and this male is the sole partner for that subject (the information on the male partner's sterility can come from the site personnel's review of the subject's medical records or interview with the subject on her medical history); male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository); male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository).
* Female subjects of childbearing potential who agree not to donate an ova during the study and for at least 30 days after the last dose of study drug.
* If male, agrees to use a condom with spermicide (note: no restrictions are required for a vasectomized male provided that his vasectomy was ≥ 4 months prior to the Screening Visit).
* Diagnosis of COPD, as defined by American Thoracic Society Global Initiative for Chronic Obstructive Lung Disease criteria
* Post-bronchodilator FEV1 ≥30% and ≤79%
* Post-bronchodilator FEV1/FVC ratio ≤70%
* Current or former smoker with a history of ≥ 10 pack-year history

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, would interfere with the subject'sability to complete the study, would interfere with the interpretation of safety or efficacy, or would present an undue risk to the subject. In cases of uncertainty, the investigator may contact the medical monitor for clarification.
* Known respiratory disorders other than COPD that, in the opinion of the investigator, may present an unacceptable safety risk to a subject's study participation or could confound the interpretation of the study safety or efficacy results. Examples include, but are not limited to: alpha-1 antitrypsin deficiency, cystic fibrosis, significant asthma, active bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, pulmonary edema, or interstitial lung disease.
* Currently taking a non-selective beta blocker. Subjects who have been on a stable dose of a cardioselective beta blocker for at least 3 months prior to screening are not excluded (examples of cardioselective beta blockers are: metoprolol, atenolol, bisoprolol, and nebivolol). Topical beta blockers for ophthalmologic conditions are permitted.
* Uncontrolled diabetes defined as HbA1c > 8.0%.
* Renal impairment defined as estimated glomerular filtration rate <50 ml/min/1.73 m2 as calculated by the Chronic Kidney Disease Epidemiology Collaboration equation.
* Liver disease as defined as one or more of the following:

  1. AST or ALT > 2 times the upper limit of normal (ULN).
  2. Total bilirubin > 2 times the ULN (subjects with bilirubin elevation patterns consistent with Gilbert's disease are permitted).
  3. A history of or suspected, in the opinion of the investigator, bleeding disorder. Subjectson therapeutic anticoagulation are not excluded if the investigator believes they are appropriately anticoagulated.
* Eosinophil count >600/mm3.
* History of a malignancy of any organ system (other than localized squamous or basal cell carcinoma of the skin) treated or untreated within the last 2 years prior to screening.
* Evidence or history of a clinically significant disease or abnormality, which, in the opinion of the investigator, would present and unacceptable safety risk to a subject's study participation or could confound the interpretation of the study efficacy or safety results. Examples of these conditions include, but are not limited to: NYHA Class II or higher congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, thyrotoxicosis, stroke, or cardiac dysrhythmia.
* Conditions which, in the opinion of the investigator, may contraindicate the use of an anticholinergic agent. Examples of these conditions may include, but are not limited to: paradoxical bronchospasm, narrow-angle glaucoma, prostatic hyperplasia, bladder neck obstruction, chronic constipation, or altered gastrointestinal motility.
* History of myasthenia gravis.
* Use of oral corticosteroids or oral antibiotics within 6 weeks prior to the Screening Visit.
* Subjects who have a positive test result on the screening urine drug screen for banned substances, including tetrahydrocannabinol or controlled substance(s) for which the subject does not have a valid prescription. Subjects taking cannabidiol should also be excluded.
* History of allergy or hypersensitivity to anticholinergic/muscarinic receptor antagonist agents, beta-2 adrenergic agonists, lactose/milk proteins, or specific intolerance to aerosolized tiotropium-containing products or known hypersensitivity to any of the proposed ingredients or components of the delivery system.
* Hospitalization for COPD or pneumonia within 8 weeks of study enrollment.
* Treatment for COPD exacerbation (defined as change in COPD symptoms requiring antibiotics and/or corticosteroids) within 12 weeks prior to enrollment.
* Have participated in pulmonary rehabilitation within 90 days of screening or are planning to participate in pulmonary rehabilitation during the course of the study
* History of 3 or more COPD exacerbations within 12 months prior to enrollment.
* Inability to refrain from COPD medications as prohibited by study protocol.
* Requires any supplemental oxygen therapy (including nocturnal oxygen).
* Acute (viral or bacterial) upper or lower respiratory tract infection, sinusitis, rhinitis, pharyngitis, urinary tract infection or illness within 6 weeks prior to enrollment.
* Abnormal and clinically significant electrocardiogram (ECG) findings, as determined by the investigator, at screening or during treatment.
* Lung volume reduction surgery within 12 months prior to the initiation of the study.
* Have an oxygen saturation <91% on room air at screening measured by pulse oximetry.
* Have participated in an investigational drug study within 30 days prior to screening. In addition, it is necessary that at least 5 half-lives of the previously administered investigational drug have elapsed by Visit 1.
* Subjects currently infected with COVID-19 or subjects who have previously been infected and have residual symptoms that, in the opinion of the investigator, would present a safety risk to study participation or could potentially interfere with the interpretation of safety or efficacy data in the current study. COVID-19 infection is defined as laboratory evidence of COVID-19 infection or by a constellation of signs/symptoms that, in the opinion of the investigator, are/were consistent with COVID-19 infection. Note: COVID-19 vaccination is not exclusionary.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Change in trough forced expiratory volume in 1 second (FEV1) compared with placebo | 22 days
  The primary outcome measure will be the change in trough FEV1 from baseline at Visit 4 in the 8 μg, 16 μg, and 24 μg doses of tiotropium bromide inhalation solution treatment groups compared with that of placebo, will be evaluated by using a mixed model for repeated measure (MMRM) in the mITT population.

SECONDARY OUTCOMES:
Change in trough FEV1 compared with placebo and Sprivia Respimat | 22 days
  The secondary outcome measure will be the change in trough FEV1 from baseline at Visit 2 and Visit 3 compared with that of placebo and from baseline at Visit 4 compared with that of Sprivia Respimat
Change in forced vital capacity (FVC) compared with placebo and Sprivia Respimat | 22 days
  The secondary outcome measure will be the change in trough forced vital capacity (FVC) from baseline at Visit 2 and Visit 3 compared with that of placebo and from baseline at Visit 4 compared with that of Sprivia Respimat

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research of Rock Hill, Rock Hill, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided